CLINICAL TRIAL: NCT01474096
Title: Effectiveness of Implementation Strategy for a Breastfeeding Guideline in Primary Care: Cluster Randomised Trial
Brief Title: Implementation Strategy for a Breastfeeding Guideline in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Susana Martín Iglesias, Nurse, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08/90680
Record Dates: First submitted 2011-11-04; First posted 2011-11-18 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Breastfeeding
Keywords: clinical practice guideline-primary health care
MeSH Terms: conditions — Breast Feeding | interventions — Lactation; Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- implementation strategy (Experimental): determining whether the use of implementation strategy (including training session, information distribution, an opinion leader) of Breastfeeding CPG in primary care is more effective than the usual practice of mere circulation.
  Interventions: Other: implementation strategy of Breastfeeding
- Conventional intervention (No Intervention)

INTERVENTIONS:
Other: implementation strategy of Breastfeeding — implementation strategy (including training session, information distribution, an opinion leader) of Breastfeeding
  Other Names: breastfeeding; clinical practice guideline; primary health care
  Arms: implementation strategy

SUMMARY:
The purpose of this study is to determine whether an implementation strategy for a breastfeeding guide is more effective than the usual practice (simple circulation of the guide) in terms of increasing the percentage of children receiving exclusive or preferential breastfeeding at 6 months age.

DETAILED DESCRIPTION:
Protection and promotion of breastfeeding is considered a priority in Europe where only 22% of children less than 6 months old are exclusively breastfed. In Spain this percentage reaches 24.8% but in our city it falls to 18.26%. Various studies emphasise that the improvement of these results falls upon the training of health professionals. Following the recommendations of a breastfeeding guide can modify professional practice and improve results with respect to patients.

Aim:to determine whether an implementation strategy for a breastfeeding guide is more effective than the usual practice (simple circulation of the guide) in terms of increasing the percentage of children receiving exclusive or preferential breastfeeding at 6 months age.

Method/Design: The present work involves a community, clinical trial, randomised by clusters in Primary Health Care Centres in Madrid Region (Spain). The project aims at determining whether the use of implementation strategy (including training session, information distribution, an opinion leader) of Breastfeeding CPG in primary care is more effective than the usual practice of mere circulation.

Number of patients required will be 240 (n=120 in the intervention group and control group), all mothers of children born during the study period (6 months), who come to the health centre on the first visit of child attention programme and give their consent to participate.

The main outcome variable is age at which breastfeeding ceases; secondary outcome variables include sex, age, educational level.

Analysis of main effectiveness will be done, comparing the proportion of patients with breastfeeding completed at 6 months in the two study groups. All statistical tests will be performed with intention to treat. Logistic regression with random effects will be used to adjust for prognostic factors. Confounding factors or factors that might alter the effect recorded will be taken into account in this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children born during the study period (6 months)
* Mothers who come to the health centre on 1st visit (child attention programme)
* Mothers who give their consent to participate.

Exclusion Criteria:

* Breastfeeding Contraindications

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
proportion of patients with breastfeeding completed at 6 months | 6 months
  Analysis of main effectiveness will be done, comparing the proportion of patients with breastfeeding completed at 6 months in the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Susana Martin, Nurse, Principal Investigator — Gerencia Atención Primaria. Madrid
Locations (1):
- Gerencia Atención Primaria, Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Gavine A, Shinwell SC, Buchanan P, Farre A, Wade A, Lynn F, Marshall J, Cumming SE, Dare S, McFadden A. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2022 Oct 25;10(10):CD001141. doi: 10.1002/14651858.CD001141.pub6. PMID 36282618
- [Derived] Martin-Iglesias S, del-Cura-Gonzalez I, Sanz-Cuesta T, Arana-Canedo Arguelles C, Rumayor-Zarzuelo M, Alvarez-de la Riva M, Lloret-Saez Bravo AM, Fernandez-Arroyo RM, Arejula-Torres JL, Aguado-Arroyo O, Gongora-Maldonado F, Garcia-Corraliza M, Sandoval-Encinas N, Tomico-delRio M, Cornejo-Gutierrez AM. Effectiveness of an implementation strategy for a breastfeeding guideline in Primary Care: cluster randomised trial. BMC Fam Pract. 2011 Dec 30;12:144. doi: 10.1186/1471-2296-12-144. PMID 22208800